CLINICAL TRIAL: NCT05907915
Title: Donor Site Healing Response to Low Level Laser Therapy Following Skin Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Mohamed Kamel, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003623
Record Dates: First submitted 2023-06-06; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2022-12

CONDITIONS: Skin Graft
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laser group (Experimental): active low level laser therapy and conventional medical treatment.
  Interventions: Device: low level laser therapy
- placebo group (Placebo Comparator): placebo laser and conventional medical treatment
  Interventions: Behavioral: placebo

INTERVENTIONS:
Device: low level laser therapy — They recieved LLLT 1 session daily, 3 session per week for 3 weeks,with the following parameters( 650 nm wavelength, 150 mw power output, 0.25 cm2 radiation area, 0.6 W/cm2 power density, continuous mode, 2 j/ cm2, 90 seconds / cm2) in addition to the conventional medical treatment and traditional wound care (dressing)
  Arms: laser group
Behavioral: placebo — They received placebo laser 1 session daily, 3 session per week for 3 weeks in addition to the conventional medical treatment and traditional wound care (dressing)
  Arms: placebo group

SUMMARY:
PURPOSE:

The purpose of the study is to evaluate the effect of (LLLT) on donor site wound healing following skin graft surgery.

BACKGROUND:

The skin graft is a beneficial reconstructive technique for accelerating wound healing .Managing donor site after graft harvesting is very important, and often, patients have more discomfort at the donor site than the recipient burn site itself.Using techniques that accelerate wound healing may enhance patient satisfaction.

Low-level laser therapy (LLLT) has been used in several medical fields, including healing of diabetic, surgical, and pressure ulcers.

Accelerating the healing process and reducing pain during healing are beneficial for the following reasons: faster return to work, lower risk of wound infection, improved quality of life, and possibly reduced need for analgesia.

HYPOTHESES:

It is hypothesized that:

Low level laser therapy has a positive effect on donor site wound healing following skin graft surgery in burned patients.

RESEARCH QUESTION:

Is low level laser therapy has a positive effect on donor site healing following skin graft surgery in burned patients?

ELIGIBILITY:
Inclusion Criteria:

* Patients are both males and females.
* Their Age will be range between 20-40 years.
* All patients suffering from third degree burn with TBSA for burn will be ranged from 20% to 35%.
* All patients undergoing split thickness skin graft surgery.
* All patients will begin the treatment program from the 1st day post operative
* All patients enrolled to the study will have their informed consent.
* All patients have donor sites from the thigh.

Exclusion Criteria:

* • Patients with associated diseases (Diabetes mellitus, infectious diseases, autoimmune disease) that will interfere with the healing process.

  * Patients taking medication that alter the healing process (e.g., corticosteroids, chemotherapy or radiation.
  * Pregnancy or epilepsy.
  * Elderly patients.
  * Subjects who have photosensitive problems
  * History of trauma or accidental injuries.
  * Skin diseases.
  * History of surgery on particular donor site.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Measurement of wound surface area at day 1 post-operative (pre-treatment)(baseline measurement) | 1 day
  Measurement of wound surface area by photography and image J software at day 1
Measurement of wound surface area at day 11 post-operative (post-treatment) | 11 day
  Measurement of wound surface area by photography and image J software at day 11
Measurement of wound surface area at day 21 post-operative (post-treatment) | 21 day
  Measurement of wound surface area by photography and image J software at day 21

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vaghardoost R, Momeni M, Kazemikhoo N, Mokmeli S, Dahmardehei M, Ansari F, Nilforoushzadeh MA, Sabr Joo P, Mey Abadi S, Naderi Gharagheshlagh S, Sassani S. Effect of low-level laser therapy on the healing process of donor site in patients with grade 3 burn ulcer after skin graft surgery (a randomized clinical trial). Lasers Med Sci. 2018 Apr;33(3):603-607. doi: 10.1007/s10103-017-2430-4. Epub 2018 Jan 24. PMID 29368069
- [Background] Assis L, Moretti AI, Abrahao TB, Cury V, Souza HP, Hamblin MR, Parizotto NA. Low-level laser therapy (808 nm) reduces inflammatory response and oxidative stress in rat tibialis anterior muscle after cryolesion. Lasers Surg Med. 2012 Nov;44(9):726-35. doi: 10.1002/lsm.22077. Epub 2012 Sep 21. PMID 23001637
- [Background] Huang J, Chen J, Xiong S, Huang J, Liu Z. The effect of low-level laser therapy on diabetic foot ulcers: A meta-analysis of randomised controlled trials. Int Wound J. 2021 Dec;18(6):763-776. doi: 10.1111/iwj.13577. Epub 2021 Mar 9. PMID 33751853
- [Background] Voineskos SH, Ayeni OA, McKnight L, Thoma A. Systematic review of skin graft donor-site dressings. Plast Reconstr Surg. 2009 Jul;124(1):298-306. doi: 10.1097/PRS.0b013e3181a8072f. PMID 19568092